CLINICAL TRIAL: NCT06622811
Title: Effect of Educational Program of Virtual Reality on Critical Thinking Disposition Among Nursing Students at Damietta University
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mona ahmed mohamed gabr, Assistant Lecturer of Nursing Administration, Faculty of Nursing, Mansoura University, Dakahlia, Egypt., Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 309
Record Dates: First submitted 2024-09-29; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Educational Program; Virtual Reality; Critical Thinking; Nursing Students

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nursing students group (Experimental): Nursing students will be scheduled to apply educational program of virtual reality to improve their critical thinking disposition.
  Interventions: Other: Students' Knowledge about Virtual Reality Questionnaire; Other: California Critical Thinking Disposition Inventory (CCTDI)

INTERVENTIONS:
Other: Students' Knowledge about Virtual Reality Questionnaire — Part I: Personal Characteristics of Nursing Students:
  It covers; age and gender.
  Part II: Students' Knowledge about Virtual Reality Questionnaire:
  This part will used to assess students' knowledge related to virtual reality that includes a definition of virtual reality, history of virtual reality, advantages and disadvantages of virtual reality on nursing education and equipment used for virtual reality and the effect virtual reality on future of education
  Scoring system:
  Respondents' answers will be scored (0) for incorrect answers, and (1) for correct answers. The overall items scores will be summed up and categorized according to the total percentages of unsatisfactory (<60%) and satisfactory (≥60%).
Other: California Critical Thinking Disposition Inventory (CCTDI) — It will consist of 24 items classify into 7 dimensions grouped as follows; truth-seeking (3 items); open-mindedness (4 items); analyticity (3 items); systematicity (4 items); critical thinking self-confidence (4 items); inquisitiveness (3 items); and cognitive maturity (3 items).
  Scoring system:
  Students asked to respond to all items with six points Likert scale as follows; strongly disagree = 1, disagree= 2, neutral = 3, sometimes agree = 4, agree = 5, and strongly agree= 6. The overall items scores will be summed up and categorized according to the total percentages of satisfactory critical thinking (≥75%) and unsatisfactory critical thinking (<75%).

SUMMARY:
The present study aims to evaluate the effect of an educational program of virtual reality on critical thinking disposition among nursing students at Damietta University.

DETAILED DESCRIPTION:
Education is the basis for a thriving society, and the transfer of knowledge has been a top priority for civilization since the very beginning, in all the world people are constantly looking for more easily, more quickly, and more effective in a world where technology is a dominant feature in our daily life.

Virtual reality in the field of medical and nursing education is defined as a type of computer-based 3D simulation that makes users feel like they are in clinical settings where they can practice skills without putting patients at risk. Therefore, such simulations with active engagement improve learning retention and enable participants to learn interactively and analyze problems.

Critical thinking disposition is one of the skills that need to be developed in the current era. Critical thinking skills can be defined as a student's ability to test their idea in dealing with problems the art of analyzing and evaluating thinking, deducting and inferring conclusions from problems and facts.

ELIGIBILITY:
Inclusion Criteria:

* Age from 21 to 22 years.
* Both sexes.
* Nursing students.

Exclusion Criteria:

- Mental retardation

Ages: 21 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 190 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Students' Knowledge about Virtual Reality Questionnaire | Two months after educational program
  Scoring system:
  Respondents' answers will be scored (0) for incorrect answers, and (1) for correct answers. The overall items scores will be summed up and categorized according to the total percentages of unsatisfactory (<60%) and satisfactory (≥60%).

SECONDARY OUTCOMES:
Students' Knowledge about Virtual Reality Questionnaire | Two months after educational program
  Scoring system:
  Students asked to respond to all items with six points Likert scale as follows; strongly disagree = 1, disagree= 2, neutral = 3, sometimes agree = 4, agree = 5, and strongly agree= 6. The overall items scores will be summed up and categorized according to the total percentages of satisfactory critical thinking (≥75%) and unsatisfactory critical thinking (<75%).

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.

REFERENCES:
- [Derived] Gabr MAM, Sleem WF, El-Wkeel NS. Effect of virtual reality educational program on critical thinking disposition among nursing students in Egypt: a quasi-experimental pretest-posttest design. BMC Nurs. 2025 Jul 7;24(1):874. doi: 10.1186/s12912-025-03488-w. PMID 40624646